CLINICAL TRIAL: NCT06263452
Title: Beta-Blocker Influences on Inflammatory and Neural Responses to Stress
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of California, Los Angeles (Other); Dartmouth College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 23-2768; 1R01HL157422-01 (NIH)
Record Dates: First submitted 2024-01-31; First posted 2024-02-16 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Disease
Keywords: Beta-Blockade; Inflammation; Neuroimaging
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation | interventions — Propranolol; Sugars

STUDY DESIGN:
Intervention Model Description: Subjects (n = 60 per condition, N = 120) will either take a one-time, 40mg dose of propranolol or an encapsulated placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double blind, randomized, placebo-controlled mechanistic clinical trial. The Investigational Drug Service will randomly assign patients to the experimental group (propranolol) or the placebo group. Research staff who have direct contact with the participant will be blind to their condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol (Experimental): Propranolol tablet, 40mg, one-time, orally
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): Encapsulated placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Tablet encapsulated to visually look identical to the placebo.
  Other Names: Inderal; Propranolol hydrochloride
  Arms: Propranolol
Drug: Placebo — Encapsulated sugar pill to visually look identical to the experimental condition.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to map the neural and molecular mechanisms underlying psychological stress-induced changes in inflammation which could reveal new targets for intervention to reduce the risk of cardiovascular disease.

DETAILED DESCRIPTION:
The proposed work will conduct a mechanistic clinical trial utilizing the non-selective beta-adrenergic receptor blocker propranolol to examine the role of beta-adrenergic signaling in shaping neural and inflammatory responses to stress. The investigators will focus on beta-adrenergic signaling given seminal pre-clinical work showing that this molecular pathway is an important driver of stress-related increases in inflammation, and initial human neuroimaging work showing that beta-blockade leads to changes in neural responses to negative stimuli. Here, the investigators will bring these two previously disparate lines of work together to determine how experimentally blocking one critical stress-signaling pathway shapes neural activity and inflammatory responses to stress. In doing so, the investigators will be advancing knowledge by mapping mechanisms (i.e., beta-adrenergic signaling), offering methodological improvements (i.e., moving beyond correlation to using pharmacological manipulations to provide causal evidence), and identifying intervention targets (i.e., the neurocognitive systems that shift activity/connectivity in response to beta-blockade). In sum, the work proposed herein is significant because it will address the mechanisms by which one critical risk factor, psychological stress, may ultimately lead to cardiovascular disease via inflammation. The proposed study also offers significant methodological improvements over past work by using neuroimaging to identify neurocognitive pathways, and pharmacology to provide causal experimental evidence to move us beyond correlation. Finally, this project is significant because it could provide insight into novel targets for future interventions.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-30 years
* Right-handed
* Fluent in English reading, writing, and speaking at least at a 10th grade level
* Body mass index (BMI) less than or equal to 35 kg/m^2

Exclusion Criteria:

Assessed as screening, reassessed at Session I:

* Non-removeable metal devices/implants/objects in the body
* Severe claustrophobia (assessed by self-report)
* Currently pregnant
* Left-handed
* Body mass index (BMI) greater than 35 kg/m^2
* History of fainting spells or any heart condition
* History of or present low resting heart rate (< 60 BPM) and/or low blood pressure (systolic blood pressure < 80mmHg)
* Self-reported physical illnesses: diabetes, cardiovascular diseases, high blood pressure, inflammatory bowel diseases, rheumatoid arthritis, asthma, autoimmune disease, Crohn's disease, ulcerative colitis, lupus
* Any self-reported diagnosed mental illness
* Current use of prescription medications (except hormonal contraceptives)
* Current or recent regular nicotine/tobacco use (cigarettes, e-cigarettes, vape, chewing tobacco, nicotine gum)
* Current regular (daily or almost daily) recreational drug use = 4 or more times per week

Instructed against during Session I, reassessed at Session II:

* Received any vaccine within the past two weeks
* Severe sleep disturbance (3-4 hours of sleep loss) the night before Session II
* Vigorous physical activity on the day of Session II
* Acute illness or allergy symptoms on the day of Session II
* Usage of over-the-counter medications on the day of Session II
* Usage of recreational drugs within 48 hours of Session II
* Usage of alcohol on the day of Session II

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in levels of pro-inflammatory cytokine interleukin-6 in response to social stress | Post-drug baseline to 90-minutes post-stress task (T-90)
  Blood plasma will be analyzed for levels of pro-inflammatory cytokine interleukin-6 (IL-6), from baseline, a baseline after drug administration, a sample 90-minutes after the stress task (T-90) measured in pg/mL. The timeline was determined on meta-analytic work showing changes in the inflammatory cytokine IL-6 are largest at 90 minutes post-stress.
Change in levels of inflammatory gene expression in response to social stress | Post-drug baseline to 30-minutes post-stress task (T-30)
  Whole blood samples will be collected in PaxGene tubes and analyzed for changes in inflammatory gene expression from baseline, a baseline after drug administration, and 30-minutes after the stress task (T-30), measured in gene transcript counts per million. The timeline is based on the Principal Investigator's work showing that changes in pro-inflammatory gene expression are observed 30-minutes post-stress.

CONTACTS AND LOCATIONS:
Overall Officials: Keely Muscatell, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Social Neuroscience and Health Laboratory, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta NK, Abrams LR, Myrskyla M. US life expectancy stalls due to cardiovascular disease, not drug deaths. Proc Natl Acad Sci U S A. 2020 Mar 31;117(13):6998-7000. doi: 10.1073/pnas.1920391117. Epub 2020 Mar 16. PMID 32179670
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Background] Lagraauw HM, Kuiper J, Bot I. Acute and chronic psychological stress as risk factors for cardiovascular disease: Insights gained from epidemiological, clinical and experimental studies. Brain Behav Immun. 2015 Nov;50:18-30. doi: 10.1016/j.bbi.2015.08.007. Epub 2015 Aug 6. PMID 26256574
- [Background] Gianaros PJ, Jennings JR. Host in the machine: A neurobiological perspective on psychological stress and cardiovascular disease. Am Psychol. 2018 Nov;73(8):1031-1044. doi: 10.1037/amp0000232. PMID 30394781
- [Background] Chida Y, Steptoe A. Greater cardiovascular responses to laboratory mental stress are associated with poor subsequent cardiovascular risk status: a meta-analysis of prospective evidence. Hypertension. 2010 Apr;55(4):1026-32. doi: 10.1161/HYPERTENSIONAHA.109.146621. Epub 2010 Mar 1. PMID 20194301
- [Background] Ginty AT, Kraynak TE, Fisher JP, Gianaros PJ. Cardiovascular and autonomic reactivity to psychological stress: Neurophysiological substrates and links to cardiovascular disease. Auton Neurosci. 2017 Nov;207:2-9. doi: 10.1016/j.autneu.2017.03.003. Epub 2017 Mar 16. PMID 28391987
- [Background] Hong S, Dimitrov S, Cheng T, Redwine L, Pruitt C, Mills PJ, Ziegler MG, Green JM, Shaikh F, Wilson K. Beta-adrenergic receptor mediated inflammation control by monocytes is associated with blood pressure and risk factors for cardiovascular disease. Brain Behav Immun. 2015 Nov;50:31-38. doi: 10.1016/j.bbi.2015.08.012. Epub 2015 Aug 20. PMID 26300225
- [Background] Devereux RB, Alderman MH. Role of preclinical cardiovascular disease in the evolution from risk factor exposure to development of morbid events. Circulation. 1993 Oct;88(4 Pt 1):1444-55. doi: 10.1161/01.cir.88.4.1444. PMID 8403291
- [Background] Black PH, Garbutt LD. Stress, inflammation and cardiovascular disease. J Psychosom Res. 2002 Jan;52(1):1-23. doi: 10.1016/s0022-3999(01)00302-6. PMID 11801260
- [Background] Ridker PM, Hennekens CH, Buring JE, Rifai N. C-reactive protein and other markers of inflammation in the prediction of cardiovascular disease in women. N Engl J Med. 2000 Mar 23;342(12):836-43. doi: 10.1056/NEJM200003233421202. PMID 10733371
- [Background] Pepys MB, Hirschfield GM, Tennent GA, Gallimore JR, Kahan MC, Bellotti V, Hawkins PN, Myers RM, Smith MD, Polara A, Cobb AJ, Ley SV, Aquilina JA, Robinson CV, Sharif I, Gray GA, Sabin CA, Jenvey MC, Kolstoe SE, Thompson D, Wood SP. Targeting C-reactive protein for the treatment of cardiovascular disease. Nature. 2006 Apr 27;440(7088):1217-21. doi: 10.1038/nature04672. PMID 16642000
- [Background] Irwin MR, Cole SW. Reciprocal regulation of the neural and innate immune systems. Nat Rev Immunol. 2011 Aug 5;11(9):625-32. doi: 10.1038/nri3042. PMID 21818124
- [Background] Flaa A, Eide IK, Kjeldsen SE, Rostrup M. Sympathoadrenal stress reactivity is a predictor of future blood pressure: an 18-year follow-up study. Hypertension. 2008 Aug;52(2):336-41. doi: 10.1161/HYPERTENSIONAHA.108.111625. Epub 2008 Jun 23. PMID 18574074
- [Background] Bosch JA, Berntson GG, Cacioppo JT, Dhabhar FS, Marucha PT. Acute stress evokes selective mobilization of T cells that differ in chemokine receptor expression: a potential pathway linking immunologic reactivity to cardiovascular disease. Brain Behav Immun. 2003 Aug;17(4):251-9. doi: 10.1016/s0889-1591(03)00054-0. PMID 12831827
- [Background] McEwen BS, Gianaros PJ. Central role of the brain in stress and adaptation: links to socioeconomic status, health, and disease. Ann N Y Acad Sci. 2010 Feb;1186:190-222. doi: 10.1111/j.1749-6632.2009.05331.x. PMID 20201874
- [Background] Gianaros PJ, Wager TD. Brain-Body Pathways Linking Psychological Stress and Physical Health. Curr Dir Psychol Sci. 2015 Aug 1;24(4):313-321. doi: 10.1177/0963721415581476. PMID 26279608
- [Background] Madden KS, Sanders VM, Felten DL. Catecholamine influences and sympathetic neural modulation of immune responsiveness. Annu Rev Pharmacol Toxicol. 1995;35:417-48. doi: 10.1146/annurev.pa.35.040195.002221. PMID 7598501
- [Background] Felten DL, Felten SY, Bellinger DL, Carlson SL, Ackerman KD, Madden KS, Olschowki JA, Livnat S. Noradrenergic sympathetic neural interactions with the immune system: structure and function. Immunol Rev. 1987 Dec;100:225-60. doi: 10.1111/j.1600-065x.1987.tb00534.x. No abstract available. PMID 3326822
- [Background] van Gool J, van Vugt H, Helle M, Aarden LA. The relation among stress, adrenalin, interleukin 6 and acute phase proteins in the rat. Clin Immunol Immunopathol. 1990 Nov;57(2):200-10. doi: 10.1016/0090-1229(90)90034-n. PMID 1698583
- [Background] Kassam KS, Mendes WB. The effects of measuring emotion: physiological reactions to emotional situations depend on whether someone is asking. PLoS One. 2013 Jun 5;8(7):e64959. doi: 10.1371/journal.pone.0064959. Print 2013. PMID 23785407
- [Background] Woo CW, Chang LJ, Lindquist MA, Wager TD. Building better biomarkers: brain models in translational neuroimaging. Nat Neurosci. 2017 Feb 23;20(3):365-377. doi: 10.1038/nn.4478. PMID 28230847
- [Background] Gianaros PJ, Sheu LK, Uyar F, Koushik J, Jennings JR, Wager TD, Singh A, Verstynen TD. A Brain Phenotype for Stressor-Evoked Blood Pressure Reactivity. J Am Heart Assoc. 2017 Aug 23;6(9):e006053. doi: 10.1161/JAHA.117.006053. PMID 28835356
- [Background] Gianaros PJ, Marsland AL, Kuan DC, Schirda BL, Jennings JR, Sheu LK, Hariri AR, Gross JJ, Manuck SB. An inflammatory pathway links atherosclerotic cardiovascular disease risk to neural activity evoked by the cognitive regulation of emotion. Biol Psychiatry. 2014 May 1;75(9):738-45. doi: 10.1016/j.biopsych.2013.10.012. Epub 2013 Oct 23. PMID 24267410
- [Background] Poldrack RA. Can cognitive processes be inferred from neuroimaging data? Trends Cogn Sci. 2006 Feb;10(2):59-63. doi: 10.1016/j.tics.2005.12.004. Epub 2006 Jan 6. PMID 16406760
- [Background] Muscatell KA, Dedovic K, Slavich GM, Jarcho MR, Breen EC, Bower JE, Irwin MR, Eisenberger NI. Greater amygdala activity and dorsomedial prefrontal-amygdala coupling are associated with enhanced inflammatory responses to stress. Brain Behav Immun. 2015 Jan;43:46-53. doi: 10.1016/j.bbi.2014.06.201. Epub 2014 Jul 9. PMID 25016200
- [Background] Fu CH, Mourao-Miranda J, Costafreda SG, Khanna A, Marquand AF, Williams SC, Brammer MJ. Pattern classification of sad facial processing: toward the development of neurobiological markers in depression. Biol Psychiatry. 2008 Apr 1;63(7):656-62. doi: 10.1016/j.biopsych.2007.08.020. Epub 2007 Oct 22. PMID 17949689
- [Background] Doehrmann O, Ghosh SS, Polli FE, Reynolds GO, Horn F, Keshavan A, Triantafyllou C, Saygin ZM, Whitfield-Gabrieli S, Hofmann SG, Pollack M, Gabrieli JD. Predicting treatment response in social anxiety disorder from functional magnetic resonance imaging. JAMA Psychiatry. 2013 Jan;70(1):87-97. doi: 10.1001/2013.jamapsychiatry.5. PMID 22945462
- [Background] van Oort J, Tendolkar I, Hermans EJ, Mulders PC, Beckmann CF, Schene AH, Fernandez G, van Eijndhoven PF. How the brain connects in response to acute stress: A review at the human brain systems level. Neurosci Biobehav Rev. 2017 Dec;83:281-297. doi: 10.1016/j.neubiorev.2017.10.015. Epub 2017 Oct 24. PMID 29074385
- [Background] Henckens MJ, van der Marel K, van der Toorn A, Pillai AG, Fernandez G, Dijkhuizen RM, Joels M. Stress-induced alterations in large-scale functional networks of the rodent brain. Neuroimage. 2015 Jan 15;105:312-22. doi: 10.1016/j.neuroimage.2014.10.037. Epub 2014 Oct 22. PMID 25462693
- [Background] Soszynski D, Kozak W, Conn CA, Rudolph K, Kluger MJ. Beta-adrenoceptor antagonists suppress elevation in body temperature and increase in plasma IL-6 in rats exposed to open field. Neuroendocrinology. 1996 May;63(5):459-67. doi: 10.1159/000127072. PMID 8738584
- [Background] Powell ND, Sloan EK, Bailey MT, Arevalo JM, Miller GE, Chen E, Kobor MS, Reader BF, Sheridan JF, Cole SW. Social stress up-regulates inflammatory gene expression in the leukocyte transcriptome via beta-adrenergic induction of myelopoiesis. Proc Natl Acad Sci U S A. 2013 Oct 8;110(41):16574-9. doi: 10.1073/pnas.1310655110. Epub 2013 Sep 23. PMID 24062448
- [Background] Johnson JD, Campisi J, Sharkey CM, Kennedy SL, Nickerson M, Greenwood BN, Fleshner M. Catecholamines mediate stress-induced increases in peripheral and central inflammatory cytokines. Neuroscience. 2005;135(4):1295-307. doi: 10.1016/j.neuroscience.2005.06.090. Epub 2005 Sep 13. PMID 16165282
- [Background] Hanke ML, Powell ND, Stiner LM, Bailey MT, Sheridan JF. Beta adrenergic blockade decreases the immunomodulatory effects of social disruption stress. Brain Behav Immun. 2012 Oct;26(7):1150-9. doi: 10.1016/j.bbi.2012.07.011. Epub 2012 Jul 24. PMID 22841997
- [Background] Hermans EJ, van Marle HJ, Ossewaarde L, Henckens MJ, Qin S, van Kesteren MT, Schoots VC, Cousijn H, Rijpkema M, Oostenveld R, Fernandez G. Stress-related noradrenergic activity prompts large-scale neural network reconfiguration. Science. 2011 Nov 25;334(6059):1151-3. doi: 10.1126/science.1209603. PMID 22116887
- [Background] Hurlemann R, Walter H, Rehme AK, Kukolja J, Santoro SC, Schmidt C, Schnell K, Musshoff F, Keysers C, Maier W, Kendrick KM, Onur OA. Human amygdala reactivity is diminished by the beta-noradrenergic antagonist propranolol. Psychol Med. 2010 Nov;40(11):1839-48. doi: 10.1017/S0033291709992376. Epub 2010 Jan 27. PMID 20102667
- [Background] von Kanel R, Kudielka BM, Metzenthin P, Helfricht S, Preckel D, Haeberli A, Stutz M, Fischer JE. Aspirin, but not propranolol, attenuates the acute stress-induced increase in circulating levels of interleukin-6: a randomized, double-blind, placebo-controlled study. Brain Behav Immun. 2008 Feb;22(2):150-7. doi: 10.1016/j.bbi.2007.07.005. Epub 2007 Sep 18. PMID 17881186
- [Background] Benschop RJ, Nieuwenhuis EE, Tromp EA, Godaert GL, Ballieux RE, van Doornen LJ. Effects of beta-adrenergic blockade on immunologic and cardiovascular changes induced by mental stress. Circulation. 1994 Feb;89(2):762-9. doi: 10.1161/01.cir.89.2.762. PMID 7508828
- [Background] O'Connor MF, Bower JE, Cho HJ, Creswell JD, Dimitrov S, Hamby ME, Hoyt MA, Martin JL, Robles TF, Sloan EK, Thomas KS, Irwin MR. To assess, to control, to exclude: effects of biobehavioral factors on circulating inflammatory markers. Brain Behav Immun. 2009 Oct;23(7):887-97. doi: 10.1016/j.bbi.2009.04.005. Epub 2009 Apr 21. PMID 19389469
- [Background] Muscatell KA, Dedovic K, Slavich GM, Jarcho MR, Breen EC, Bower JE, Irwin MR, Eisenberger NI. Neural mechanisms linking social status and inflammatory responses to social stress. Soc Cogn Affect Neurosci. 2016 Jun;11(6):915-22. doi: 10.1093/scan/nsw025. Epub 2016 Mar 15. PMID 26979965
- [Background] Eisenberger NI, Inagaki TK, Muscatell KA, Byrne Haltom KE, Leary MR. The neural sociometer: brain mechanisms underlying state self-esteem. J Cogn Neurosci. 2011 Nov;23(11):3448-55. doi: 10.1162/jocn_a_00027. Epub 2011 Mar 31. PMID 21452934
- [Background] Muscatell KA, Moieni M, Inagaki TK, Dutcher JM, Jevtic I, Breen EC, Irwin MR, Eisenberger NI. Exposure to an inflammatory challenge enhances neural sensitivity to negative and positive social feedback. Brain Behav Immun. 2016 Oct;57:21-29. doi: 10.1016/j.bbi.2016.03.022. Epub 2016 Mar 28. PMID 27032568
- [Background] Kemeny ME. Psychobiological responses to social threat: evolution of a psychological model in psychoneuroimmunology. Brain Behav Immun. 2009 Jan;23(1):1-9. doi: 10.1016/j.bbi.2008.08.008. Epub 2008 Sep 10. PMID 18809488
- [Background] Dickerson SS, Kemeny ME. Acute stressors and cortisol responses: a theoretical integration and synthesis of laboratory research. Psychol Bull. 2004 May;130(3):355-91. doi: 10.1037/0033-2909.130.3.355. PMID 15122924
- [Background] Dickerson SS, Gable SL, Irwin MR, Aziz N, Kemeny ME. Social-evaluative threat and proinflammatory cytokine regulation: an experimental laboratory investigation. Psychol Sci. 2009 Oct;20(10):1237-44. doi: 10.1111/j.1467-9280.2009.02437.x. Epub 2009 Sep 14. PMID 19754527
- [Background] Wager TD, Waugh CE, Lindquist M, Noll DC, Fredrickson BL, Taylor SF. Brain mediators of cardiovascular responses to social threat: part I: Reciprocal dorsal and ventral sub-regions of the medial prefrontal cortex and heart-rate reactivity. Neuroimage. 2009 Sep;47(3):821-35. doi: 10.1016/j.neuroimage.2009.05.043. Epub 2009 May 22. PMID 19465137
- [Background] Dickerson SS, Mycek PJ, Zaldivar F. Negative social evaluation, but not mere social presence, elicits cortisol responses to a laboratory stressor task. Health Psychol. 2008 Jan;27(1):116-21. doi: 10.1037/0278-6133.27.1.116. PMID 18230022
- [Background] Slavich GM, Way BM, Eisenberger NI, Taylor SE. Neural sensitivity to social rejection is associated with inflammatory responses to social stress. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14817-22. doi: 10.1073/pnas.1009164107. Epub 2010 Aug 2. PMID 20679216
- [Background] Marsland AL, Walsh C, Lockwood K, John-Henderson NA. The effects of acute psychological stress on circulating and stimulated inflammatory markers: A systematic review and meta-analysis. Brain Behav Immun. 2017 Aug;64:208-219. doi: 10.1016/j.bbi.2017.01.011. Epub 2017 Jan 12. PMID 28089638
- [Background] Rohleder N. Stimulation of systemic low-grade inflammation by psychosocial stress. Psychosom Med. 2014 Apr;76(3):181-9. doi: 10.1097/PSY.0000000000000049. PMID 24608036
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Steptoe A, Hamer M, Chida Y. The effects of acute psychological stress on circulating inflammatory factors in humans: a review and meta-analysis. Brain Behav Immun. 2007 Oct;21(7):901-12. doi: 10.1016/j.bbi.2007.03.011. Epub 2007 May 1. PMID 17475444
- [Background] Jolink TA, Fendinger NJ, Alvarez GM, Feldman MJ, Gaudier-Diaz MM, Muscatell KA. Inflammatory reactivity to the influenza vaccine is associated with changes in automatic social behavior. Brain Behav Immun. 2022 Jan;99:339-349. doi: 10.1016/j.bbi.2021.10.019. Epub 2021 Nov 5. PMID 34748895
- [Background] Fredrickson BL, Grewen KM, Coffey KA, Algoe SB, Firestine AM, Arevalo JM, Ma J, Cole SW. A functional genomic perspective on human well-being. Proc Natl Acad Sci U S A. 2013 Aug 13;110(33):13684-9. doi: 10.1073/pnas.1305419110. Epub 2013 Jul 29. PMID 23898182
- [Background] Fredrickson BL, Grewen KM, Algoe SB, Firestine AM, Arevalo JM, Ma J, Cole SW. Psychological well-being and the human conserved transcriptional response to adversity. PLoS One. 2015 Mar 26;10(3):e0121839. doi: 10.1371/journal.pone.0121839. eCollection 2015. PMID 25811656
- [Background] Dawkins L, Corcoran O. Acute electronic cigarette use: nicotine delivery and subjective effects in regular users. Psychopharmacology (Berl). 2014 Jan;231(2):401-7. doi: 10.1007/s00213-013-3249-8. Epub 2013 Aug 27. PMID 23978909
- [Background] Cosme D, Zeithamova D, Stice E, Berkman ET. Multivariate neural signatures for health neuroscience: assessing spontaneous regulation during food choice. Soc Cogn Affect Neurosci. 2020 Nov 10;15(10):1120-1134. doi: 10.1093/scan/nsaa002. PMID 31993654
- [Background] Sporns O. Graph theory methods: applications in brain networks. Dialogues Clin Neurosci. 2018 Jun;20(2):111-121. doi: 10.31887/DCNS.2018.20.2/osporns. PMID 30250388
- [Background] Steptoe A, Ronaldson A, Kostich K, Lazzarino AI, Urbanova L, Carvalho LA. The effect of beta-adrenergic blockade on inflammatory and cardiovascular responses to acute mental stress. Brain Behav Immun. 2018 May;70:369-375. doi: 10.1016/j.bbi.2018.03.027. Epub 2018 Mar 26. PMID 29588232